CLINICAL TRIAL: NCT00224666
Title: Evaluation of the Effectiveness of Stimulation Cortex Sensorimotor for the Treatment of Rebel Neuropathic Pains
Brief Title: Efficacy of Cortex Stimulation in Neuropathic Pain
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: P000901; AOM98134
Record Dates: First submitted 2005-09-16; First posted 2005-09-23 (Estimated); Last update posted 2007-01-11 (Estimated); Status verified 2007-01

CONDITIONS: Rebel Neuropathic Pains
Keywords: Cortex stimulation ,Rebel neuropathic pains

INTERVENTIONS:
Device: Cortex stimulation

SUMMARY:
The pains chronic neurogeneses remain difficult to treat whatever are their origin and their localization. The pharmacological therapeutic arsenal answers only partially the symptomatology often very invalidating which these chronic painful patients present. Electric stimulations of the central nervous system currently validated, in particular of the posterior cords of marrow made a significant improvement in a certain number of indications. Nevertheless, considerable patients are not relieved significantly, in particular those presenting of the pains neurogeneses of central origin (syndromes thalamic for example). It is within this framework that recently the stimulation of the sensorimotor cortex developed.

Principal objective: evaluation of the technique of stimulation under cortical on neuropathic pains .

DETAILED DESCRIPTION:
The pains chronic neurogeneses remain difficult to treat whatever are their origin and their localization. The pharmacological therapeutic arsenal answers only partially the symptomatology often very invalidating which these chronic painful patients present. Electric stimulations of the central nervous system currently validated, in particular of the posterior cords of marrow made a significant improvement in a certain number of indications. Nevertheless, considerable patients are not relieved significantly, in particular those presenting of the pains neurogeneses of central origin (syndromes thalamic for example). It is within this framework that recently the stimulation of the sensorimotor cortex developed.

ELIGIBILITY:
Inclusion Criteria:

* Neurofibromatosis,
* Rebel chronic neuropathic pain with duration > 1 year and AVS > = 4

Exclusion Criteria:

* Cancer
* Epilepsy
* Cognitive deterioration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16
Dates: Start 2001-03; Study Completion 2005-11

PRIMARY OUTCOMES:
Efficacy of 50% of EVS at 3 weeks

SECONDARY OUTCOMES:
Efficacy of 50% of EVS at 6 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: N'GUYEN, Pr,MD,PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hopital Henri Mondor, Créteil, France

REFERENCES:
- [Background] Drouot X, Oshino S, Jarraya B, Besret L, Kishima H, Remy P, Dauguet J, Lefaucheur JP, Dolle F, Conde F, Bottlaender M, Peschanski M, Keravel Y, Hantraye P, Palfi S. Functional recovery in a primate model of Parkinson's disease following motor cortex stimulation. Neuron. 2004 Dec 2;44(5):769-78. doi: 10.1016/j.neuron.2004.11.023. PMID 15572109
- [Background] Lefaucheur JP, Drouot X, Menard-Lefaucheur I, Zerah F, Bendib B, Cesaro P, Keravel Y, Nguyen JP. Neurogenic pain relief by repetitive transcranial magnetic cortical stimulation depends on the origin and the site of pain. J Neurol Neurosurg Psychiatry. 2004 Apr;75(4):612-6. doi: 10.1136/jnnp.2003.022236. PMID 15026508